CLINICAL TRIAL: NCT05391854
Title: Clinical Study to Assess the Long-term Effect of Pep2Dia® on Glucose Homeostasis in Prediabetic Subjects: a 12-week Randomized, Multicenter, Double-blind, Placebo-controlled, Parallel Study
Brief Title: Clinical Study to Assess the Long-term Effect of Pep2Dia® on Glucose Homeostasis in Prediabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ingredia S.A. (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BTS1777/21
Record Dates: First submitted 2022-05-06; First posted 2022-05-26 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pep2dia (Active Comparator)
  Interventions: Dietary Supplement: Pep2dia
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pep2dia — 700 mg Pep2Dia® 15 min prior to breakfast and 700 mg Pep2Dia® 15 min prior to dinner
  Arms: Pep2dia
Dietary Supplement: Placebo — 700 mg placebo 15 min prior to breakfast and 700 mg placebo 15 min prior to dinner
  Arms: Placebo

SUMMARY:
The goal is to assess the long-term effect of Pep2Dia® compared to placebo intake on blood glucose homeostasis. Respective improvements will be assessed by changes in glycated haemoglobin (HbA1c) before and after the 12-weeks intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects (minimum one third of each gender) with prediabetic HbA1c values between 5.7% and 6.4% and/or fasting glucose ≥ 5.6 mmol/L (≥ 100 mg/dL) and < 7.0 mmol/L (< 125 mg/dL) (in venous plasma) (twice confirmed at two independent days if HbA1c is < 5.7%)
* Age: 25-70 years
* Body mass index 19-35 kg/m2
* Current Non-smoker
* Availability and presence in the study units for approx. 3.5 hours/ week for 2 times.
* Signed informed consent form
* No changes in food habits or physical activity 3 months prior to screening and during the study
* If applicable, stable intake of chronic medication of at least 4 weeks

Exclusion Criteria:

* Subjects with diagnosed Type 2-Diabetes with medical treatment
* Presence of disease or drug(s) influencing digestion and absorption of nutrients
* Intake of medications known to affect glucose tolerance, e.g., diabetic medication SGLT-2 inhibitors, GLP-1 receptor agonists, steroids, protease inhibitors or antipsychotics
* Chronic intake of substances affecting blood coagulation (e.g. acetylic acid (100 mg as standard prophylactic treatment allowed when dose is stable 1 month prior to screening), anticoagulants, diuretics, thiazides (diuretics and thiazides allowed e.g. for hypertension treatment when dose is stable 1 month prior to screening)), which in the Investigator's opinion would impact patient safety
* Severe liver or renal disease or laboratory evidence of hepatic dysfunction (i.e. alkaline phosphatase, ALT, AST >3 x ULN)
* Acute gastrointestinal diseases including diarrhea and/or vomiting within the last 2 weeks
* Known inflammatory or malignant gastrointestinal diseases (i.e. colitis ulcerosa, Morbus Crohn, celiac disease, malignant diseases e.g. colon-cancer, rectum cancer, pancreatitis)
* Clinically relevant findings as established by medical history, physical examination, clinical laboratory and/or vital signs
* Major medical or surgical event requiring hospitalization within the previous 3 months
* Intake of food supplements known to affect glucose tolerance, e.g., cinnamon capsules, conjugated linoleic acids, omega-3 fatty acids
* Intake of antibiotics within 4 weeks before the test days
* Known alcohol abuse or drug abuse
* Pregnant or breast-feeding women
* Weight loss intervention or recent body weight change >5 kg during last 3 months
* Known or suspected allergy to any component of the investigational product(s) (e.g. milk protein)
* Blood donation within 4 weeks prior to Visit 1 or during the study
* Anticipating any planned changes in lifestyle for the duration of the study
* Participation in another clinical intervention study within the last 4 weeks and concurrent participation in another intervention clinical study
* Subject unable to co-operate adequately

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) | Before treatment (baseline = day 0); at the end of the treatment (after 3 months = day 85)
  Change from baseline Glycated haemoglobin (HbA1c) at 3 months

SECONDARY OUTCOMES:
Glucose-iAUC(0-180min) | Day 1; Day 85
  Area under the curve calculated as the incremental area under the blood glucose response curve, ignoring the area beneath the fasting concentration
Cmax | Day 1; Day 85
  Maximum blood glucose concentration
Delta Cmax | Day 1; Day 85
  Maximum increase of glucose (Cmax minus baseline value)
Tmax | Day 1; Day 85
  Time to reach maximum blood glucose concentration
Tbaseline | Day 1; Day 85
  First time to reach baseline again after increase or decrease in blood glucose
ISI 0-120min | Day 1; Day 85
hsCRP | Day 1; Day 85
GLP-1 | Day 1; Day 85
Body composition measurement | Day 1; Day 85
  Evaluation of the fat mass/lean mass ratio by bioelectrical impedance analysis
SF-12 (Short-fom 12) | Day 1; Day 85
  Score from 12 to 60. Higher score mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotesys, Esslingen am Neckar, Germany